CLINICAL TRIAL: NCT01727765
Title: Inspiratory Muscle Training as a Novel Approach in the Treatment of Asthma
Brief Title: Inspiratory Muscle Training and Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Mitch Lomax, Senior Lecturer, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMT and Asthma
Record Dates: First submitted 2012-11-07; First posted 2012-11-16 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Asthma, inspiratory muscle training
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): 6 weeks of inspiratory muscle training, 6 days per week. The intensity of training will be equivalent to up to 50% of pre-training maximal inspiratory mouth pressure and will be adapted weekly to reflect the improvement in inspiratory muscle strength
  Interventions: Other: inspiratory muscle training
- Sham Comparator (Sham Comparator): 6 weeks of sham inspiratory muscle training, 6 days per week. The intensity of training will be equivalent to 5% of pre-training inspiratory mouth pressure throughout the 6 week period.
  Interventions: Other: inspiratory muscle training

INTERVENTIONS:
Other: inspiratory muscle training — Both groups will undertake six weeks of inspiratory muscle training (POWERbreathe, H&B International Ltd, UK), six days per week, with the only difference being the load set on the inspiratory muscle training device. For the real inspiratory muscle training group this load will be set to around 50% of maximal inspiratory mouth pressure and for the sham inspiratory muscle training group this load will be set to around 5% of maximal inspiratory mouth pressure.

SUMMARY:
This is a pilot study which will assess the feasibility of a follow on main study. This study will examine the impact of inspiratory muscle training on quality of life, rescue drug medication usage, and other markers of asthma in adult asthmatics in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Asthma Control Questionnaire score of ≥ 1.5
* 10 mg or less of prednisolone (or equivalent) daily
* Aged 18 to 59 years inclusive
* Able to provide written informed consent

Exclusion Criteria:

* Any significant heart or lung disease other than asthma including any previous history of pneumothorax
* Patients with a concomitant condition (including clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease) not controlled with treatment, making implementation of the protocol or interpretation of the study results difficult
* Women who are pregnant
* Forced expiratory volume in one second of less than 50% best or predicted
* A history of smoking 20 cigarettes a day for 20 years or more (or an equivalent amount)
* Undertaken a structured program of inspiratory muscle training within the past three months
* Currently a participant in another interventional study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Respiratory Centre, Queen Alexandra Hospital, Cosham, Portsmouth, Hampshire
  - University of Portsmouth, Portsmouth, Hampshire

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Sham Comparator
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Sham Comparator | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12) | 54 (14) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximal Inspiratory Mouth Pressure (MIP)
Description: MIP is a surrogate measure of inspiratory muscle strength and was measured pre and post 6 weeks of either experimental or sham inspiratory muscle trianing (IMT).
Time Frame: pre (after the 4 week run-in) and post 6 weeks of IMT
Population: As this was a feasibility study, statistical analysis was not required
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Experimental: Undertook 6 weeks of real IMT
- Sham: undertook 6 weeks of sham IMT
Arm/Group | Experimental | Sham
Number analyzed (Participants) | 8 | 8
kPa
  MIP pre training | 9.36 (2.63) | 9.37 (2.90)
  MIP post training | 10.55 (2.72) | 9.21 (2.66)

ADVERSE EVENTS:
Time Frame: 12 weeks. This encompassed the 4 week run-in period, 2 weeks for testing (one week pre IMT and 1 week post IMT) and 6 weeks for IMT.
Arm/Group | Experimental | Sham Comparator
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes